CLINICAL TRIAL: NCT05828290
Title: The Effect of the Little Yogis do Yoga Program on Sleeping Habits in Pre-school Children: Randomized Controlled Trial
Brief Title: The Effect of Yoga on Gaining Sleep Habits in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayşegül İşler Dalgıç, Prof., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAEK-34
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Yoga; Preschool Children; Sleep Habit

STUDY DESIGN:
Intervention Model Description: pretest, posttest design, follow-up, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: At the end of the research, the groups will be coded as "A" and "B". Statistical analysis will be made by the statistics expert who is blinded to the groups in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): The "Little Yogis Doing Yoga" Program was started to be implemented by the researcher for 4 weeks, 2 days a week for 30 minutes, separately for each group, in a way to form 2 groups.
  Interventions: Behavioral: Child Yoga
- Control Group (No Intervention): Children in the control group will continue their routine education at school.

INTERVENTIONS:
Behavioral: Child Yoga — The children's yoga consists of compositions such as playing, stories, postures, breathing exercises, imitations things in nature, memory games, music, dance and daydreaming.
  Arms: Yoga Group

SUMMARY:
This study was planned to determine the effect of the "Little Yogis Doing Yoga" Program, which will be created within the scope of the research, on getting children aged 5-6 years old to sleep habits. This study was planned in a pretest, posttest design, follow-up, randomized controlled study. The sample of the study will consist of 36 children (18 children in the intervention group, 18 children in the control group) in the 5-6 age group in Antalya between 15 March and 15 June 2023. The "Little Yogis Doing Yoga" Program, which was created within the scope of the research, will be applied to the children in the intervention group in two groups, two days a week, for 4 weeks, 30 minutes each, by the researcher who received child yoga specialization training. Data will be collected with Child and Family Information Form and Child Sleep Habits Questionnaire-CSHQ). CSHQ, T0-Pretest (Before the Program "Little Yogis Doing Yoga"), T1-Interim follow-up (after the program ends) and T2-Posttest (1 month after the program is completed) will be filled by the parents. Statistical Package for the Social Sciences (SPSS) 24.0 package program will be used in the analysis of the data.

DETAILED DESCRIPTION:
Preschool (three-six years) is a period in which the physical, psychomotor, social-emotional, cognitive and language development of the child is completed to a large extent. In this period when the growth-development process is very important, healthy and regular sleep plays an active role in many developmental areas of children, especially in brain development. For this reason, examining and arranging the sleep habits of children in the preschool period is of great importance for the healthy completion of the process. The aim of this study is to determine the sleep habits of children in the 5-6 age group and to determine the effect of children's yoga on these habits. This study was planned to determine the effect of the "Little Yogis Doing Yoga" Program, which will be created within the scope of the research, on instilling sleep habits in children aged 5-6 years.

ELIGIBILITY:
Inclusion Criteria:

* 5-6 years old
* No school attendance problems
* Those who have the cognitive ability to carry out the commands given during child yoga.
* Having no physical problems that may prevent active participation in children's yoga
* Children who do not have an obstacle to communication (sight, hearing problems, etc.) and whose parents' consent to participate in the study are approved

Exclusion Criteria:

* Children who are actively attending any children's yoga program

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Children's Sleep Habits Questionnaire (CSHQ) | CSHQ score will evaluate at baseline
  To gain children the ability to sleep habits. The Children's Sleep Habits Questionnaire (CSHQ)- Abbreviated Form developed by Owens et al. consists of 33 items in total. In the scale, bedtime resistance (1,3,4,5,6,8 items), delay in falling asleep (2nd item), sleep duration (9,10,11 items), sleep anxiety (5,7,8, 21st items), night awakenings (items 16,24,25), parasomnias (12,13,14,15,17,22,23), disruption of breathing during sleep (items 18,19,20), day Eight subscales were defined as sleepiness (items 26,27,28,29,30,31,32,33). A total of 41 points is considered the cutoff point, and values above this are considered 'clinically significant'.
Children's Sleep Habits Questionnaire (CSHQ) | CSHQ score will evaluate one month later
  To gain children the ability to sleep habits. The Children's Sleep Habits Questionnaire (CSHQ)- Abbreviated Form developed by Owens et al. consists of 33 items in total. In the scale, bedtime resistance (1,3,4,5,6,8 items), delay in falling asleep (2nd item), sleep duration (9,10,11 items), sleep anxiety (5,7,8, 21st items), night awakenings (items 16,24,25), parasomnias (12,13,14,15,17,22,23), disruption of breathing during sleep (items 18,19,20), day Eight subscales were defined as sleepiness (items 26,27,28,29,30,31,32,33). A total of 41 points is considered the cutoff point, and values above this are considered 'clinically significant'.
Children's Sleep Habits Questionnaire (CSHQ) | CSHQ score will evaluate two month later
  To gain children the ability to sleep habits. The Children's Sleep Habits Questionnaire (CSHQ)- Abbreviated Form developed by Owens et al. consists of 33 items in total. In the scale, bedtime resistance (1,3,4,5,6,8 items), delay in falling asleep (2nd item), sleep duration (9,10,11 items), sleep anxiety (5,7,8, 21st items), night awakenings (items 16,24,25), parasomnias (12,13,14,15,17,22,23), disruption of breathing during sleep (items 18,19,20), day Eight subscales were defined as sleepiness (items 26,27,28,29,30,31,32,33). A total of 41 points is considered the cutoff point, and values above this are considered 'clinically significant'.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Nur Ünver, RN, Study Chair — Akdeniz University
Locations (1):
- Aysegul ISLER DALGIC, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No